CLINICAL TRIAL: NCT06670339
Title: Effect of Pre-cooling the Body on Whole-body Heat Exchange in Young Males During Exercise in the Heat
Brief Title: Effect of Pre-cooling on Whole-body Heat Loss During Exercise-heat Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Professor, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HEPRU-2024-08-B
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Thermoregulation; Cold Exposure; Heat Stress; Exercise
Keywords: Cold Stress; Heat Stress; Heat Dissipation; Physical Activity; Performance; Athletes; Workers
MeSH Terms: conditions — Heat Stress Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Cooling (Active Comparator): Participants will complete 60 min of continuous semi-recumbent cycling at a fixed metabolic heat load (200 W/m2) in the heat (wet-bulb globe temperature of 29°C; 37.5°C and 35% relative humidity) (Control condition) without pre-cooling.
  Interventions: Other: No Cooling
- Pre-Cooling (Experimental): Participants will undergo a cold-water immersion (~17°C) to elicit a decrease in rectal temperature by 0.5°C from baseline values. Thereafter, once the target temperature is achieved, participants will complete 60 min of continuous moderate-intensity cycling (200 W/m2) in the heat (wet-bulb globe temperature of 29°C; 37.5°C and 35% relative humidity).
  Interventions: Other: Pre-Cooling

INTERVENTIONS:
Other: No Cooling — Participants will not be pre-cooled prior to completing a 60-minute moderate-intensity exercise bout in the heat.
  Arms: No Cooling
Other: Pre-Cooling — Participants will be immersed in cold (~17°C) water to elicit a decrease in rectal temperature by 0.5°C from baseline values prior to completing a 60-min moderate-intensity exercise bout in the heat.
  Arms: Pre-Cooling

SUMMARY:
Endurance exercise performance declines in hot environments as core body temperature increases. To enhance performance, body pre-cooling strategies, such as cold-water immersion have been employed to lower resting core temperature thereby increasing the body's heat storage capacity. In turn, the increase in body core temperature associated with exercise in the heat is blunted, allowing the individual to exercise at higher intensity and or for a longer period of time. However, the mechanisms by which pre-cooling impacts heat exchange during exercise remain unclear. While existing research has focused on the performance benefits of pre-cooling the body, relatively little is known about the impacts of pre-cooling on whole-body heat exchange during an exercise-heat stress. Investigators will therefore evaluate whole-body heat exchange (dry ± evaporative heat loss as assessed using a direct air calorimeter) during a prolonged (1-hour) moderate-intensity cycling bout in the heat (wet-bulb globe temperature of 29°C; equivalent to 37.5°C, 35% relative humidity) performed with and without pre-cooling by cool-water (~17°C) immersion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young males (18-30 years)
* Non-smoking
* English or French speaking
* Ability to provide informed consent

Exclusion Criteria:

* Presence of chronic diseases (e.g., hypertension, diabetes)
* Acute illness (e.g., flu, COVID-19)
* Physical restriction limiting physical activity
* Use of medication judged by the patient or investigators to make participation in this study inadvisable.
* Sedentary

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Evaporative heat loss at end exercise | Final 15 minutes of the 60 minutes exercise bout
  Evaporative heat loss as assessed using a direct air calorimeter
Dry heat loss at end exercise | Final 15 minutes of the 60 minutes exercise bout
  Total dry heat loss as assessed using a direct air calorimeter
Total heal loss at end exercise | Final 15 minutes of the 60 minutes exercise bout
  Net heat loss (dry plus/minus evaporative heat exchange) as assessed using a direct air calorimeter
Body heat storage during the 60-minute exercise bout | Over the 60 minute exercise bout
  Change in body heat storage (i.e., amount of heat stored in the body) calculated as the temporal summation of metabolic heat production and total heat loss
Core temperature at end of exercise | Final 15 minutes of exercise
  Rectal temperature during final 15 minutes of exercise. Rectal temperature is measured continuously throughout the intervention.
Relative change in core temperature at end of exercise | Change over the 60-minute exercise bout
  Change in rectal temperature from baseline resting.
Heart rate at end exercise | Final 15 minutes of exercise
  Heart rate during final 15 minutes of exercise. Rectal temperature is measured continuously throughout the intervention.
Mean skin temperature at end of exercise | Final 15 minutes of exercise
  Skin temperature measured continuously at 4-sites (chest, upper arm, thigh, calf) with mean value calculated as weighted value of 4 sites - upper arm, 30%; chest, 30%; thigh, 20%; and calf, 20%
Relative change in skin temperature at end of exercise | Change over the 60-minute exercise bout
  Change in skin temperature from baseline resting as assessed at 4-sites (chest, upper arm, thigh, calf) with mean value calculated as weighted value of 4 sites - uper arm, 30%; chest, 30%; thigh, 20%; and calf, 20%
Thermal sensation A at end exercise | Final 15 minutes of exercise
  Thermal sensation assessed via a self-report questionnaire upon verbal prompting (7-point scale; -3: cold to +3: hot)
Thermal sensation B at end exercise | Final 15 minutes of exercise
  Thermal sensation assessed via a self-report questionnaire upon verbal prompting (7-point scale; 0: neutral to 7: extremely hot)
Thermal comfort at end exercise | Final 15 minutes of exercise
  Thermal comfort assessed via a self-report questionnaire upon verbal prompting (4-point scale; 1: comfortable to 4: very uncomfortable)
Thirst sensation at end exercise | Final 15 minutes of exercise
  Thirst sensation assessed via a self-report questionnaire upon verbal prompting (9-point scale; 1: not thirsty at all to 9: very, very thirsty)
Rating of perceived exertion | Final 15 minutes of exercise
  Perceived exertion assessed via a self-report questionnaire upon verbal prompting (6: no exertion at all to 20: maximal exertion)

SECONDARY OUTCOMES:
Heart rate variability at end of exercise | Final 15 minutes of exercise
  Measures of variability computed from the time, frequency, time-frequency, scale-invariant, entropy, and other nonlinear domains (R-R interval data extracted from the electrocardiogram). Measured continuously using a holter monitor with Zymed placement

CONTACTS AND LOCATIONS:
Overall Officials: Glen P Kenny, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available with approved analysis plan and signed access agreement
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Following publication of the main study report(s)
Access Criteria: Approved analysis plan and signed access agreement